CLINICAL TRIAL: NCT03280758
Title: Effects of Muscle Strength Training on Glycemic Control, Muscle Mass, Muscle Strength and Functional Capacity in Older Adults With Type II Diabetes: A Randomised Controlled Trial
Brief Title: Muscle Strength Training for Older Adults With Type II Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Resistance training; Diabetes Mellitus; blood-glucose control; Muscle; Function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not know the intervention of each subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle strengthening group (Experimental): Participants will be required to perform muscle strengthening exercises 3 hours per week. Close kinetic chain exercises will be performed progressively according to the ACSM guidelines over the 4-month intervention period. The exercise intervention will be conducted by an experienced sports trainer.
  Interventions: Behavioral: Muscle Strengthening exercises
- Control group (No Intervention): No exercise training.

INTERVENTIONS:
Behavioral: Muscle Strengthening exercises — Participants will be required to participate in resistance training 3 hours per week.
  Arms: Muscle strengthening group

SUMMARY:
This randomised controlled trial aims to investigate a resistance training program for improving glycemic control, muscle mass, strength and functional performance in older patients with Type II Diabetes (T2 DM).

60 subjects will be randomly allocated to either a muscle strengthening group or a no exercise control group.

Muscle strengthening group will receive resistance training 3 times per week (1 hour/session).

The control group will not receive any training but can continue usual medical care and daily activities.

Primary outcomes: glycemic control and lipid profile Secondary outcomes: muscle mass and strength, and functional capacity Data will be collected at baseline (pre-test) and after a 4-month intervention (post-test).

DETAILED DESCRIPTION:
This study aims to investigate a resistance training program for improving glycemic control, muscle mass, strength and functional performance in older patients with Type II Diabetes (T2 DM).

This is a single-blinded, randomized controlled trial. 60 subjects will be randomly allocated to either a muscle strengthening group or a no exercise control group.

Information on demographic characteristics, body composition, muscle strength, functional capacity and glycemic control will be collected at baseline (pre-test) and after a 4-month intervention (post-test). Muscle strengthening group will receive resistance training 3 times per week (1 hour/session).

The control group will not receive any training but can continue usual medical care and daily activities.

ELIGIBILITY:
Inclusion Criteria:

* T2 DM
* 60-75 years old
* ability to perform exercise

Exclusion Criteria:

* Advanced hypertension (≥ 160/100 mm Hg)
* severe obesity (BMI ≥ 48kg/m2)
* insulin pump user
* coronary heart disease history
* chronic obstructive pulmonary disease
* advanced neuropathy
* learning or mental disorder, or
* any other diseases that prevent subjects from exercising safely.
* Those who participate in regular resistance or aerobic exercises will also be excluded.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose level | 4 months
Lipid profiles | 4 months
  HDL, LDL, Trig

SECONDARY OUTCOMES:
Muscle strength | 4 months
  Whole body
Muscle mass | 4 months
  Whole body
Functional performance | 4 months
  Walking ability

CONTACTS AND LOCATIONS:
Overall Officials: Siu Ming Fong, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nolan CJ, Damm P, Prentki M. Type 2 diabetes across generations: from pathophysiology to prevention and management. Lancet. 2011 Jul 9;378(9786):169-81. doi: 10.1016/S0140-6736(11)60614-4. Epub 2011 Jun 24. PMID 21705072
- [Background] Leenders M, Verdijk LB, van der Hoeven L, Adam JJ, van Kranenburg J, Nilwik R, van Loon LJ. Patients with type 2 diabetes show a greater decline in muscle mass, muscle strength, and functional capacity with aging. J Am Med Dir Assoc. 2013 Aug;14(8):585-92. doi: 10.1016/j.jamda.2013.02.006. Epub 2013 Mar 26. PMID 23537893
- [Background] Shishikura K, Tanimoto K, Sakai S, Tanimoto Y, Terasaki J, Hanafusa T. Association between skeletal muscle mass and insulin secretion in patients with type 2 diabetes mellitus. Endocr J. 2014;61(3):281-7. doi: 10.1507/endocrj.ej13-0375. Epub 2014 Jan 10. PMID 24420336
- [Background] Dunstan DW, Daly RM, Owen N, Jolley D, De Courten M, Shaw J, Zimmet P. High-intensity resistance training improves glycemic control in older patients with type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1729-36. doi: 10.2337/diacare.25.10.1729. PMID 12351469
- [Background] American Diabetes Association. Diabetes mellitus and exercise. Diabetes Care. 2000 Jan;23 Suppl 1:S50-4. No abstract available. PMID 12017678
- [Background] Albright A, Franz M, Hornsby G, Kriska A, Marrero D, Ullrich I, Verity LS. American College of Sports Medicine position stand. Exercise and type 2 diabetes. Med Sci Sports Exerc. 2000 Jul;32(7):1345-60. doi: 10.1097/00005768-200007000-00024. PMID 10912903
- [Background] Black LE, Swan PD, Alvar BA. Effects of intensity and volume on insulin sensitivity during acute bouts of resistance training. J Strength Cond Res. 2010 Apr;24(4):1109-16. doi: 10.1519/JSC.0b013e3181cbab6d. PMID 20093961
- [Background] Baldi JC, Snowling N. Resistance training improves glycaemic control in obese type 2 diabetic men. Int J Sports Med. 2003 Aug;24(6):419-23. doi: 10.1055/s-2003-41173. PMID 12905089